CLINICAL TRIAL: NCT07370259
Title: The Effect of Training Provided Through Gamification Method on the Menstruation and Genital Hygiene Behaviors of Female Students
Brief Title: Gamification Method on the Menstruation and Genital Hygiene Behaviors of Female Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lokman Hekim University (Other Government)
Responsible Party: Principal Investigator, Özlem Ülkü BULUT, Assistant Profesor, Lokman Hekim University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: genital hijyen
Record Dates: First submitted 2026-01-18; First posted 2026-01-27 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Menstrual Hygiene; Genital Hygiene Behaviors; Adolescent Health; Health Education; Gamification
Keywords: Adolescent Health; Gamification; Genital Hygiene; Menstrual Hygiene
MeSH Terms: conditions — Health Education

STUDY DESIGN:
Intervention Model Description: The study was planned as a one-group pretest-posttest quasi-experimental study so as to evaluate the effect of gamification method on menstruation and genital hygiene behaviors of female students.
Masking Description: his study was conducted as a one-group pretest-posttest quasi-experimental design without any masking procedure. Participants and investigators were aware of the intervention since the educational program was delivered through an interactive, web-based gamified platform. Outcome assessments were based on self-reported questionnaires administered before and one month after the training. No blinding was feasible due to the educational nature of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gamified Training Group (Experimental): All participants received the web-based gamified educational program designed to improve menstruation and genital hygiene behaviors. The program included four interactive online sessions of approximately 20 minutes each, incorporating gamification elements such as avatars, badges, levels, and virtual rewards to enhance engagement. Pre- and post-test assessments were administered to evaluate changes in hygiene behaviors.
  Interventions: Behavioral: Gamified Training Program

INTERVENTIONS:
Behavioral: Gamified Training Program — The intervention consisted of a web-based gamified educational program developed using Web 2.0 tools. The program included four interactive online sessions, each lasting approximately 20 minutes, and aimed to improve menstruation and genital hygiene behaviors among female students. Gamification elements such as avatars, badges, levels, and virtual rewards were integrated following the D6 design model (Discover, Define, Design, Develop, Deploy, Determine). The training combined visuals, videos, and quizzes to enhance engagement and motivation. Post-intervention assessments were conducted one month after the completion of all sessions to evaluate behavioral outcomes.

SUMMARY:
This quasi-experimental study aimed to evaluate the effect of a gamification-based educational intervention on menstruation and genital hygiene behaviors among female students. The study was conducted with 77 female students aged 10-15 years who were attending a public secondary school in Ankara, Türkiye, during the 2023-2024 academic year. The intervention consisted of a web-based gamified education program developed by the researchers using Web 2.0 tools and implemented through an interactive online platform in four sessions. Data were collected before and one month after the intervention using the Menstrual Hygiene Behaviors Form and the Genital Hygiene Behaviors Scale (GHBS). Findings indicated a significant improvement in general hygiene, menstrual hygiene, and awareness of abnormal findings after the intervention (p < 0.05). The study suggests that gamified online education can be an effective and engaging approach to improving menstrual and genital hygiene behaviors among adolescent girls.

DETAILED DESCRIPTION:
This study was designed as a one-group pretest-posttest quasi-experimental research to evaluate the effect of a gamification-based educational intervention on menstruation and genital hygiene behaviors among female students. The research was carried out with 77 female students aged 10-15 years who were attending a public secondary school in Ankara, Türkiye, during the 2023-2024 academic year. Participants were recruited on a voluntary basis, and written informed consent was obtained from their parents prior to participation.

The intervention consisted of a web-based gamified educational program developed by the researchers using Web 2.0 tools. The content was structured based on the D6 gamification design model (Discover, Define, Design, Develop, Deploy, Determine). The educational material was delivered in four interactive online sessions, each lasting approximately 20 minutes. The sessions included visual materials, short videos, quizzes, badges, levels, and virtual rewards to increase motivation and engagement. The educational modules covered reproductive anatomy, the importance of hand and personal hygiene, perineal hygiene, the use of menstrual hygiene products, and waste management.

Data were collected using the Menstrual Hygiene Behaviors Form and the Genital Hygiene Behaviors Scale (GHBS), which evaluates three dimensions: general hygiene, menstrual hygiene, and awareness of abnormal findings. Measurements were obtained before and one month after the intervention.

Statistical analyses were performed using SPSS version 27. Paired-sample t-tests and Wilcoxon tests were used to compare pretest and posttest results. A statistically significant improvement was observed in students' general hygiene, menstrual hygiene, and awareness of abnormal findings scores after the gamified education program (p < 0.05).

The study received ethical approval from the Lokman Hekim University Non-Interventional Research Ethics Committee (Protocol No: 2023/01-45; Date: February 28, 2023). Institutional permission was also obtained from the Ankara Provincial Directorate of the Ministry of National Education.

Overall, the findings suggest that gamified online education can effectively improve menstrual and genital hygiene behaviors among adolescent girls. Integrating gamification-based approaches into school health education programs may contribute to sustainable hygiene behaviors and promote adolescent health.

ELIGIBILITY:
Inclusion Criteria:

* Female students enrolled in a public secondary school in Ankara
* Aged between 10 and 15 years
* Having experienced menarche (menstruating)
* Able to read and understand Turkish
* Having internet access to complete online training
* Willing to participate voluntarily in the study
* Parental written consent provided

Exclusion Criteria:

* Students who have not yet experienced menarche
* Incomplete questionnaire or missing data
* Lack of parental consent
* Students who did not complete all four gamified education sessions
* Students with any condition limiting participation in online learning activities

Ages: 10 Years to 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 77 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Change in Genital Hygiene Behaviors Scale (GHBS) Total Score | From baseline (pre-test) to 1 month after completion of the gamified educational program
  The Genital Hygiene Behavior Scale (GHBS) is a 23-item Likert-type instrument designed to assess genital hygiene behaviors across three subdomains: general hygiene, menstrual hygiene, and awareness of abnormal genital findings. Each item is scored on a 5-point Likert scale, yielding a total score ranging from 23 to 115, with higher scores indicating better genital hygiene behaviors.

SECONDARY OUTCOMES:
Change in General Hygiene Subscale Score (GHBS) | Baseline to 1 month post-intervention
  Evaluates basic hygiene practices such as handwashing, perineal cleaning, and drying habits. The General Hygiene subscale consists of 12 items scored on a 5-point Likert scale. Subscale scores range from 12 to 60, with higher scores indicating better general genital hygiene behaviors.
Change in Menstrual Hygiene Subscale Score (GHBS) | Baseline to 1 month post-intervention
  Assesses menstrual hygiene management practices such as product use, cleaning, and waste disposal. The Menstrual Hygiene subscale consists of 8 items scored on a 5-point Likert scale. Subscale scores range from 8 to 40, with higher scores indicating better menstrual hygiene behaviors.
Change in Awareness of Abnormal Findings Subscale Score (GHBS) | Baseline to 1 month post-intervention
  Measures students' awareness of symptoms indicating possible infection or abnormal genital conditions. The Awareness of Abnormal Findings subscale consists of 3 items scored on a 5-point Likert scale. Subscale scores range from 3 to 15, with higher scores indicating greater awareness of abnormal genital findings.
Change in Menstrual Hygiene Behaviors Form Score | Baseline to 1 month post-intervention
  Menstrual Hygiene Behaviors Form: It was developed by the researchers based on the literature and consists of 4 categorical items assessing bathing style, cleaning method, genital cleansing direction, and drying practices during menstruation. The items are evaluated individually, and no total score is calculated

CONTACTS AND LOCATIONS:
Overall Officials: Ozlem Ulku Bulut, Assistant Professor, Study Chair — Lokman Hekim University
Locations (1):
- Lokman Hekim University Etlik Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study involved minors and was conducted under strict ethical confidentiality agreements. Only aggregate (summary) data will be reported in publications.